CLINICAL TRIAL: NCT03258749
Title: Efficiency of Twice Daily Formoterol Versus Once Daily Tiotropium in Patients With GOLD A/B COPD: a Randomised, Open-label, Multicentre Trial
Brief Title: Efficiency of Twice Daily Formoterol Versus Once Daily Tiotropium in Patients With GOLD A/B COPD
Acronym: FACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Shengqing Li, Chief Physician,Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2017-009
Record Dates: First submitted 2017-08-13; First posted 2017-08-23 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; GOLD; formoterol; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Formoterol (Active Comparator): inhaled formoterol(4.5μg, bid)
  Interventions: Drug: Formoterol
- Tiotropium (Experimental): inhaled Tiotropium(18μg, qd)
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium — inhaled Tiotropium(18μg, qd)
  Arms: Tiotropium
Drug: Formoterol — inhaled formoterol(4.5μg, bid)
  Arms: Formoterol

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a disease state characterized by persistent airflow limitation and associated with an accelerated decline in lung function, impaired quality of life, hospitalization, and increased mortality. As a major public health problem, COPD is predicted to rank as the fifth burden of diseases in the world by 2020. Thus, prevention of exacerbations is a important goal in the management of COPD. The Global Initiative for Chronic Obstructive Lung Disease (GOLD) Scientific Committee launched a joint project in 1998. Its goals were to raise awareness of COPD and to improve prevention and treatment of COPD patients around the world. In the 2017 GOLD guidelines, inhaled long-acting bronchodilators, including inhaled long-acting muscarinic antagonists (LAMAs) and inhaled long-acting beta-agonists (LABAs), are recommended for the management of all stable COPD patients. However, it is not known whether LABA or LAMA will be more effective for initial relief of symptoms in patients with GOLD A/B COPD. In this multicenter, randomized study, the investigators evaluate the efficacy of formoterol(LABA) and tiotropium(LAMA) in the treatment of patients with GOLD A/B COPD. The primary endpoint is postbronchodilator FEV1, and the secondary endpoints include the frequency of COPD exacerbation, other lung function parameters, CCQ score and mMRC/CAT score.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of group A or group B stable COPD. Must be able to inhale Formoterol or Tiotropium.

Exclusion Criteria:

Asthma. Cystic fibrosis. Bronchiectasis. Lung cancer. Glaucoma. Tachyarrhythmia or other serious heart diseases. Prostatic hyperplasia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
postbronchodilator FEV1 | 12 months
  a post-bronchodilator forced expiratory volume in one second

SECONDARY OUTCOMES:
the frequency of COPD exacerbation | 12 months
  the frequency of COPD exacerbation
other lung function parameters | 12 months
  other lung function parameters(%FEV1, FEV1/FVC)
CCQ score | 12 months
  Clinical COPD Questionnaire score
mMRC score | 12 months
  modified Medical Research Council score
CAT score | 12 months
  COPD Assessment Test score

CONTACTS AND LOCATIONS:
Overall Officials: Shengqing Li, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan hospital,Fudan university, Shanghai, Shanghai Municipality, China